CLINICAL TRIAL: NCT06107998
Title: Comparison of the Audible Leak-balloon Palpation Method and the Stethoscope-guided Method for Endotracheal Tube Cuff Inflation
Brief Title: Comparison of Different Methods for Determining Endotracheal Cuff Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mustafa Soner Ozcan, Assistant professor, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SNR-10/143
Record Dates: First submitted 2023-10-21; First posted 2023-10-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Anesthesia, General; Intubation, Intratracheal
Keywords: Cuff pressure; Endotracheal intubation; endotracheal tube; inflation; measurement
MeSH Terms: interventions — Stethoscopes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the person who intubates the patient and inflates the cuff using a method will know what the procedure is.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stethoscope (Experimental): Patients whose endotracheal tube cuff is inflated via a stethoscope
  Interventions: Other: stethoscope
- Audible leak/Balloon palpation (Active Comparator): Patients whose endotracheal tube cuff is inflated via audible leak/balloon palpation method.
  Interventions: Other: Audible leak/Balloon palpation

INTERVENTIONS:
Other: stethoscope — endotracheal tube cuff will be inflated via stethoscope guidance
  Arms: Stethoscope
Other: Audible leak/Balloon palpation — endotracheal tube cuff will be inflated via audible leak/balloon palpation method
  Arms: Audible leak/Balloon palpation

SUMMARY:
The goal of this clinical trial is to test whether the stethoscope can be used as a method of assessing endotracheal cuff pressure as effectively as a manometer and also to compare it with the balloon palpation/audible leak method frequently used in clinical practice in adult patients undergoing general anesthesia.

The main questions it aims to answer are:

* Is the stethoscope as effective as a manometer in assessing endotracheal cuff pressure?
* Is there a difference between stethoscope and audible leak/balloon palpation methods in assessing endotracheal cuff pressure? Participants will be randomly divided into 2 groups.
* Group P: After intubation, endotracheal cuff pressure will be assessed by audible leak/balloon palpation.
* Group S: After intubation, endotracheal cuff pressure will be assessed with a stethoscope.
* Control will be carried out with a manometer and the pressure values obtained in the groups will be corrected.

Researchers will compare ''stethoscope'' and ''audible leak/balloon palpation'' groups to see if which method is effective like a manometer.

DETAILED DESCRIPTION:
Although the use of a manometer is recommended in daily practice to evaluate endotracheal tube cuff pressure for intubated patients, the cuff is still inflated using balloon palpation or audible leakage methods in many centers. Manometers may not be available in most centers. An acceptable cuff pressure ranges from 20 to 30 cm H2O. While the risk of aspiration increases below 20 cm H2O, at values above 30 cm H2O the circulation of the tracheal mucosa begins to deteriorate and related complications like ulceration, stenosis, and even fistula may develop.

The authors hypothesize that the stethoscope is as effective as a manometer in assessing endotracheal tube cuff pressure where a manometer is not available.

After informed consent is obtained from patients who meet the inclusion criteria for the study, the patients will be intubated following anesthesia induction and the method by which the patients' endotracheal tube cuffs will be inflated will be determined in a randomized manner using the sealed envelope method. Then, the cuff pressures will be checked with a manometer by an expert who does not know the method by which the cuff is inflated, if necessary, it will be corrected and the data will be recorded with the code assigned to the method. Statistical evaluations will be made on the data obtained by an analyst who does not know the names of the methods and which method was applied to which patient.

The difference between our study and previous studies:

* Previous studies had small numbers of patients.
* The authors designed a randomized controlled study with triple masking.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Planning the operation under general anesthesia
* Performing endotracheal intubation during general anesthesia
* Elective surgeries
* Volunteering to participate in the study

Exclusion Criteria:

* Having a history of difficult intubation before
* Difficulty during intubation (repeated intubation attempts, etc.)
* rapid sequence intubation requirement
* Planning to undergo head and neck surgery
* Those with tracheal stenosis
* Previous intervention to the neck area (radiotherapy, tracheotomy, etc.)
* Pregnancy
* Obesity
* Those with respiratory diseases (COPD, asthma, etc.)
* Emergency surgery
* American Society of Anaesthesiologists physical status>3
* Refusing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
cuff pressure of air introduced | After the patients are intubated and tube cuff inflated
  After the cuffs inflated using the specified methods are checked with a manometer, it will be noted whether there is any difference between the required pressures (centimeter of water/cm H2O).
cuff volume of air introduced | After the patients are intubated and tube cuff inflated
  After the cuffs inflated using the specified methods are checked with a manometer, it will be noted whether there is any difference between the required additional volumes (milliliters/mL).

SECONDARY OUTCOMES:
endotracheal tube diameters | After induction of anesthesia and intubation
  The authors will also investigate whether cuff pressure adjustments vary by endotracheal tube diameter (Millimeter/mm)
endotracheal tube brands | After induction of anesthesia and intubation
  The authors will also investigate whether cuff pressure adjustments vary by endotracheal tube brands. The brands will be noted as A, B, C, D..etc.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Soner Özcan, M.D., Principal Investigator — Suleyman Demirel University,Faculty of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Suleyman Demirel University, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is finished, data from the study will be shared when reasonable reasons are presented.

REFERENCES:
- [Background] Kumar CM, Seet E, Van Zundert TCRV. Measuring endotracheal tube intracuff pressure: no room for complacency. J Clin Monit Comput. 2021 Feb;35(1):3-10. doi: 10.1007/s10877-020-00501-2. Epub 2020 Mar 20. PMID 32198671
- [Background] Duarte NMDC, Caetano AMM, Arouca GO, Ferrreira AT, Figueiredo JL. [Subjective method for tracheal tube cuff inflation: performance of anesthesiology residents and staff anesthesiologists. Prospective observational study]. Braz J Anesthesiol. 2020 Jan-Feb;70(1):9-14. doi: 10.1016/j.bjan.2019.09.010. Epub 2020 Feb 19. PMID 32199655
- [Result] Borhazowal R, Harde M, Bhadade R, Dave S, Aswar SG. Comparison between Two Endotracheal Tube Cuff Inflation Methods; Just-Seal Vs. Stethoscope-Guided. J Clin Diagn Res. 2017 Jun;11(6):UC01-UC03. doi: 10.7860/JCDR/2017/26301.10017. Epub 2017 Jun 1. PMID 28764268
- [Result] Satya Prakash MVS, Aravind C, Mohan VK. Comparative evaluation of three methods of endotracheal tube cuff inflation for adequacy of seal. J Anaesthesiol Clin Pharmacol. 2022 Oct-Dec;38(4):588-593. doi: 10.4103/joacp.JOACP_560_20. Epub 2022 Jun 15. PMID 36778817
- [Result] Unsal O, Seyhun N, Turk B, Ekici M, Dobrucali H, Turgut S. The Evaluation of Upper Airway Complications Secondary to Intubation: Cuff Pressure Manometer Versus Conventional Palpation Method. Sisli Etfal Hastan Tip Bul. 2018 Dec 28;52(4):289-295. doi: 10.5350/SEMB.20171214085933. eCollection 2018. PMID 32774093